CLINICAL TRIAL: NCT06608836
Title: Acute Effects of Cryotherapy on Muscle Mechanical Properties and Muscle Activation Changes
Brief Title: Acute Effects of Cryotherapy on Muscle Properties
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, Gamze Aydin, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulOkanUni
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Cryotherapy Effect
Keywords: cryotherapy; muscles; acute effect; muscle strength; electromyography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): An ice massage will be applied to the quadrices muscle for a duration of 3 minutes.
  Interventions: Other: an ice massage
- Group 2 (Experimental): A cold spray application will be performed to the quadrices muscle.
  Interventions: Other: the cold spray

INTERVENTIONS:
Other: an ice massage — an ice massage
  Arms: Group 1
Other: the cold spray — the cold spray
  Arms: Group 2

SUMMARY:
The main aim of this study is to investigate the acute effects of cryotherapy on muscle mechanical properties, muscle strength, and activation changes in healthy subjects.

DETAILED DESCRIPTION:
What changes occur in muscle stiffness following cryotherapy application? How does cryotherapy affect muscle strength? How does cryotherapy impact muscle activation? Are there differences in muscle mechanical properties, muscle strength, and muscle activation between different cryotherapy methods (ice massage and cold spray)? How do the effects of cryotherapy on muscle mechanical properties, muscle strength, and muscle activation change over time?

ELIGIBILITY:
Inclusion Criteria:

* Being willing to participate in the study
* Being between the ages of 18 and 35

Exclusion Criteria:

* Having undergone orthopedic surgery involving the lower extremity

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
myoton pro device | 3 months
  elasticity of muscle will assess by myoton pro device
muscle strength | 3 months
  muscle strength will assess by dynanometer
electromyography device | 3 months
  activation of quadriceps muscle will assess by electromyography device

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Aydın, PhD, Principal Investigator — Okan University

IPD SHARING:
Plan to Share IPD: No